CLINICAL TRIAL: NCT02085954
Title: Evaluation of a Training in the Walking With Exosquelette
Acronym: LOKOMAT
Status: Completed | Type: Observational
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Principal Investigator, Nicolas ROCHE, MD, Centre d'Investigation Clinique et Technologique 805
Other Study IDs: 12077
Record Dates: First submitted 2014-01-28; First posted 2014-03-13 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2015-10

CONDITIONS: Gait; Stroke; Robotic Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Stroke patients in the investigators rehabilitation unit follow gait trainings with robotic-assistive devices such as Lokomat. Patients able to walk alone are also assessed with 3D gait analysis. The objective of this study is to assess the effects of gait training in Lokomat on biomecanic gait parameters in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* single stroke
* able to walk alone
* > 18years

Exclusion Criteria:

* Cognitive impairments disturbing understanding
* Uncontrolled medical disorder associated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stroke patients follow in our rehabilitation hospital, able to walk alone
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
peak knee flexion (degrees) | participants will be followed for the duration of hospital stay, an expected average of 1 week

SECONDARY OUTCOMES:
hip and ankle kinematics (degrees) | participants will be followed for the duration of hospital stay, an expected average of 1 week
kinetics (newton/meter) | participants will be followed for the duration of hospital stay, an expected average of 1 week
spatio temporal parameter (m/s) | participants will be followed for the duration of hospital stay, an expected average of 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Raymond Poincare, Garches, Garches, France